CLINICAL TRIAL: NCT00458809
Title: A Phase I Evaluation of Intraperitoneal Hyperthermic Chemoperfusion With Oxaliplatin for Peritoneal Surface Disemmination of Appendiceal and Colorectal Cancer
Brief Title: Intraperitoneal Hyperthermic Perfusion With Oxaliplatin in Treating Patients With Stage IV Peritoneal Cancer Due to Appendix Cancer or Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540283; P30CA012197 (NIH); CCCWFU-59106; CCCWFU-IRB00000847; CCCWFU-59106 IPHC
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma of the Appendix; Colorectal Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; carcinoma of the appendix; recurrent rectal cancer; stage IV rectal cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hyperthermic Chemoperfusion with Oxaliplatin 200 mg/m2 (Experimental): Intraperitoneal Hyperthermic Chemoperfusion with Oxaliplatin 200 mg/m2
  Interventions: Drug: oxaliplatin
- Hyperthermic Chemoperfusion with Oxaliplatin 250 mg/m2 (Experimental): Intraperitoneal Hyperthermic Chemoperfusion with Oxaliplatin 250 mg/m2
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — Intraperitoneal Hyperthermic Chemoperfusion with Oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hyperthermia therapy kills tumor cells by heating them to several degrees above normal body temperature. Adding chemotherapy to hyperthermia and infusing it directly into the abdomen may kill more tumor cells. Giving this treatment after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I trial is studying the side effects and best dose of intraperitoneal hyperthermic perfusion with oxaliplatin in treating patients with stage IV peritoneal cancer due to appendix cancer or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of intraperitoneal hyperthermic chemoperfusion with oxaliplatin in patients with stage IV peritoneal surface malignancies from primary colorectal or appendiceal cancer.
* Determine the pharmacokinetics of this drug in perfusate, normal peritoneum, and peritoneal surface tumors in these patients.
* Evaluate the expression of proteins involved in the apoptotic and stress-inducible heat shock protein pathways (e.g., Fas, TRAIL, DISC components [FADD, TRADD, FLIP, and caspase 8], mitochondrial proteins [Bax, Bak, Bcl-2, Bcl-X_L], and heat shock proteins [HSPs 27, 40, 70 and 90]) before and after drug therapy.

OUTLINE: This is a nonrandomized, open-label, dose-escalation study.

Patients undergo gross tumor resection on day 1. After tumor debulking, patients receive oxaliplatin over 2 hours by intraperitoneal hyperthermic chemotherapy (IPHC).

Cohorts of 3-6 patients in each stratum receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients undergo blood and tissue sampling before and after IPHC for pharmacokinetic studies and for evaluation of proteins involved in apoptosis and heat-shock-mediated cell death (e.g., Fas, TRAIL, FADD, TRADD, FLIP, caspase 8, Bax, Bak, Bcl-X, and heat shock proteins 27, 40, 70, and 90).

After completion of study treatment, patients are followed periodically for at least 1 year.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal or appendiceal cancer

  * Stage IV disease
  * Peritoneal surface dissemination of disease (peritoneal carcinomatosis)
* Measurable disease according to RECIST criteria
* No active CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* No active infection or fever ≥ 101.3°F within the past 3 days
* No other malignancy within the past 5 years except curatively treated basal cell skin cancer, cervical intra-epithelial neoplasia, or localized prostate cancer with a current prostate-specific antigen of < 1.0 mg/dL on 2 successive evaluations, ≥ 3 months apart, with the last evaluation within the past 4 weeks
* No peripheral neuropathy ≥ grade 2
* No other medical condition, mental illness, or substance abuse that, in the opinion of the principal investigator, would preclude study compliance
* No known hypersensitivity to any component of oxaliplatin
* No known HIV positivity
* No hepatitis B or C positivity (active, previously treated, or both)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients and their partners must use effective contraception during and for 90 days after completion of study treatment

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery, radiotherapy, and other anticancer therapies
* More than 30 days since prior and no other concurrent investigational therapy
* No prior radiotherapy to > 25% of bone marrow
* No prior allogeneic stem cell transplantation
* No concurrent antiretroviral therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 18 days
  Maximum tolerated dose will be determined by the absence of dose limiting toxicites (serious adverse events related to Oxaplatin dosing within 18 days of administration)

SECONDARY OUTCOMES:
Pharmacokinetics | day of surgery (day one)
  Evaluation of the pharmacokinetics of oxaliplatin in perfusate, normal peritoneum, and peritoneal surface tumors during intraperitoneal hyperthermic chemoperfusion
Change in the phenotypic expression of proteins involved in the apoptotic and heat-stress inducible pathways | Day of surgery (day one)
  Analysis of the expression of proteins involved in the apoptotic and stress-inducible heat shock protein pathways before and after intraperitoneal hyperthermic chemoperfusion with oxaliplatin. These proteins shall include cellular levels of Fas and TRAIL, components of the DISC (FADD, TRADD, FLIP, and Caspase 8), mitochondrial proteins (Bax, Bak, Bcl-2, and Bcl-XL), and the heat shock protein family (HSPs 27, 40, 70, and 90).

CONTACTS AND LOCATIONS:
Overall Officials: John H. Stewart, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Stewart JH 4th, Shen P, Russell G, Fenstermaker J, McWilliams L, Coldrun FM, Levine KE, Jones BT, Levine EA. A phase I trial of oxaliplatin for intraperitoneal hyperthermic chemoperfusion for the treatment of peritoneal surface dissemination from colorectal and appendiceal cancers. Ann Surg Oncol. 2008 Aug;15(8):2137-45. doi: 10.1245/s10434-008-9967-1. Epub 2008 May 21. PMID 18493824